CLINICAL TRIAL: NCT04131062
Title: Randomized Trial to Determine Whether eConsent is Non-Inferior to Standard Consent Among Prospective Biobank Participants
Brief Title: Trial to Compare eConsent With Standard Consent Among Prospective Biobank Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Michelle N. Meyer, Assistant Professor, Geisinger Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2017-0334; R01CA211723-03S1 (NIH)
Record Dates: First submitted 2019-10-10; First posted 2019-10-18 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Lynch Syndrome
Keywords: Inherited conditions; Biobank enrollment
MeSH Terms: conditions — Colorectal Neoplasms, Hereditary Nonpolyposis

STUDY DESIGN:
Intervention Model Description: One control arm (traditional, human-mediated consent) compared against one intervention arm (electronic-based consent using the Sage eConsent framework).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (no intervention) (No Intervention): Consented using the traditional, human-mediated consent process already in use for MyCode consenting.
- Electronic Consent (iPad) (Experimental): Consented using the Sage eConsent framework, which presents participants with an iPad that describes MyCode and allows participants to choose to learn more information at various steps along the process.
  Interventions: Behavioral: Electronic Consent (iPad)

INTERVENTIONS:
Behavioral: Electronic Consent (iPad) — Participants who receive the intervention will be consented using an electronic app presented via iPad and developed according to the Sage eConsent framework.
  Arms: Electronic Consent (iPad)

SUMMARY:
The goal of this trial is to determine whether the Sage eConsent framework (presented using an electronic application) is non-inferior to traditional, paper-based, human-mediated consent-and therefore could be part of an acceptable population screening approach to identifying patients and others with actionable hereditary syndromes-and to increase basic knowledge about patients' informational needs about different aspects of genetic/omic screening. After receiving either 1) the traditional consenting approach, or 2) a consenting approach presented on an electronic tablet, the investigators will test for differences between these two arms in a variety of outcome measures including objective and perceived comprehension, time spent and informational needs, and enrollment decision, among others.

DETAILED DESCRIPTION:
The usual consent process for MyCode proceeds as follows: each day, trained MyCode consenters receive a list of patients who are eligible to be approached about MyCode and are scheduled to be seen that day in certain clinics in Geisinger's two-state catchment area. (Any Geisinger patient is eligible who has not previously enrolled in, or declined to enroll in, MyCode.) When an eligible patient arrives at the clinic, the consenter approaches them, confirms their identity, and then asks them if they would like to hear about MyCode. If they decline, the consenter thanks the patient for their time and the encounter is over. If the patient agrees, the consenter goes through a script that the MyCode team has developed from the written consent form that highlights the most important aspects of MyCode, including return of actionable results to participants and their primary care physicians, genetic privacy, and data sharing for research purposes. At the end of the script, the consenter invites and answers questions from the patient. Next, the consenter hands the patient the 7-page written consent form and asks if they would like a few minutes to review it. Finally, the consenter asks the patient whether they wish to enroll in MyCode or not and records their answer-Yes, No, or Thinking (i.e., the patient needs more time to consider)-into the patient's electronic health record.

In the present trial, patients are randomized at the individual level to receive either this usual consent or eConsent via iPad app. During the pilot phase of this trial, 11 Research Assistants (RAs) were trained on both MyCode consenting and on this trial's protocol. As per usual care, the RAs receive a daily list of MyCode-eligible patients scheduled to appear in clinic. And, as per usual care, the RAs approach the patient, confirm their identity, and ask if they wish to learn about MyCode. Those who do are then randomized to the usual care (paper) or eConsent (iPad) arm of the trial, according to whether the current time, as indicated by digital stopwatches, ends in an even or odd number. In the paper arm, the consent process proceeds as usual, with only two minor changes: 1) the RA uses the stopwatch to time the duration of the consent encounter (beginning from the moment they are randomized to the paper arm and ending when either the consent process is interrupted-e.g., because the patient is called back to the examination room-or when the consent process terminates with an enrollment decision (Yes, No, or Thinking); and 2) the RA uses a tracking sheet to record MyCode response rate (i.e., patients approached who did not want to hear about MyCode) and study attrition (e.g., consent process was interrupted). In the iPad arm, the RA hands the patient the iPad and explains that the interactive app will tell them all about MyCode. Patients reluctant to use an iPad are encouraged once to try, with the RA showing them that all that is involved is tapping, but patients who continue to resist are switched to the paper arm and this is noted on the tracking sheet. In the iPad arm, the RA also records whether the patient asks the RA any questions about MyCode and, as with the paper arm, when a patient declines to hear about MyCode and when the consent process is interrupted.

In both arms, patients are then asked to complete a survey, which serves as the primary source of data for the study. The survey is administered on paper in the paper arm and on iPad (via the Qualtrics platform) in the iPad arm. The eConsent app generates a random study ID number that is sent to Qualtrics, where the user's click behavior during the consent process (e.g., time spent on each screen and in total, whether the user clicked "learn more" on each page, (in)correct answers to teach-back questions) is anonymously combined with their survey responses. Survey questions are closed-end (true/false, multiple choice, Likert scale) and based on the Quality of Informed Consent and All of Us participant-provided information surveys.

This study is designed to be powered at 99% to detect an effect of modest size (half a point on the comprehension quiz), requiring 526 participants. Very high levels of power (here, 95% or 99%)-as opposed to the more standard benchmark power level of 80%-are desirable in tests of non-inferiority so that investigators can be as certain as possible that an inference of "no effect" is not a Type II error. In the very unlikely event that data collection proceeds much more slowly than it has in the pilot, the study retains 95% power to detect a one-half question effect with only 372 participants.

ELIGIBILITY:
Inclusion Criteria:

* None

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 703 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-05-19 (Actual); Study Completion 2022-05-19 (Actual)

PRIMARY OUTCOMES:
Mean objective comprehension: eConsent vs. control | Immediately after consent decision
  Objective comprehension quiz score measured using 10-item quiz (minimum = 0; maximum = 10; higher scores indicate greater comprehension)
Mean perceived comprehension: eConsent vs. control | Immediately after consent decision
  Subjective, self-reported comprehension measures using 8-item survey (minimum on each item = 1; maximum = 4; higher scores indicate greater perceived comprehension)
Mean perceived duration of consent process: eConsent vs. control | Immediately after consent decision
  Survey (1 item) (minimum on item = 1; maximum = 4; higher scores indicate shorter perceived duration)
Mean perceived ease of consent process: eConsent vs. control | Immediately after consent decision
  (minimum on item = 1; maximum = 4; higher scores indicate greater perceived ease)
Item-specific objective comprehension | Immediately after consent decision
  Item-specific responses to comprehension quiz (10 items) (six multiple choice items with four options each; four true/false items)
Item-specific perceived comprehension | Immediately after consent decision
  Item-specific perceived comprehension (8 items) (minimum on each item = 1; maximum = 4; higher scores indicate greater perceived comprehension)
Time spent considering each element of MyCode | Measured during consent
  In-app click behavior (time spent per screen) (continuous measure of time in seconds; greater values indicate more time spent)
Expressed informational needs for each element of MyCode | Measured during consent
  In-app click behavior (rate of choosing to "learn more" per element) (more clicks indicate greater expressed informational needs)
Sociodemographic variables | Immediately after consent decision
  Sociodemographic survey (17 items including discrete and continuous measure; "select all that apply" questions; and the ability to "prefer not to answer")
Actual duration of consent process | Measured during consent
  Measured using stopwatch (paper arm) or app (iPad arm). Greater numbers indicate longer duration.
MyCode enrollment decision | Immediately after consent process
  Survey (1 item) (measured as "yes," "no," or "thinking (needs more time)"

CONTACTS AND LOCATIONS:
Overall Officials: Michelle N Meyer, PhD, JD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD (none of which includes identifiers) will be de-identified and shared. We will consider whether certain demographic variables need to be blurred to prevent identification of participants.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be shared no later than publication of results, and will be available indefinitely.
Access Criteria: The data will be available to anyone for general research use. It will be shared at CT.gov, Open Science Framework (OSF), or both.

REFERENCES:
- [Derived] Vogt-Yerem RL, Heck PR, Gjorgjieva T, Mestechkin R, Rosica D, Huynh A, Chabris CF, Kirchner HL, Wilbanks J, Doerr M, Wagner JK, Meyer MN. eConsent vs. Traditional Consent Among Prospective Biobank Participants: A Randomized Trial. medRxiv [Preprint]. 2025 Nov 2:2025.10.30.25339179. doi: 10.1101/2025.10.30.25339179. PMID 41282898